CLINICAL TRIAL: NCT04310319
Title: Wishing to Decrease Aquaresis in ADPKD Patients Treated With a V2Ra; the Effect of Regulating Protein and Salt
Acronym: WATER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Esther Meijer (Other)
Responsible Party: Sponsor-Investigator, Esther Meijer, Principal Investigator, nephrologist, University Medical Center Groningen
Organization: University Medical Center Groningen (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: NL2019WATER
Record Dates: First submitted 2020-03-03; First posted 2020-03-17 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Polycystic Kidney, Autosomal Dominant; ADPKD; Autosomal Dominant Polycystic Kidney
Keywords: ADPKD; aquaresis; Vasopressine V2 receptor antagonist; Diet
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant | interventions — Proteins; Salts

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Normal salt, low protein treatment period (Other): 6 grams of sodium chloride daily / Placebo
  Interventions: Dietary Supplement: Sodiumchloride; Dietary Supplement: Placebo comparator (protein)
- Normal salt, normal protein treatment period (Other): 6 grams of sodium chloride daily / 40 grams of protein daily
  Interventions: Dietary Supplement: Sodiumchloride; Dietary Supplement: Protein
- Low salt, low protein treatment period (Other): Double placebo
  Interventions: Dietary Supplement: Placebo comparator (salt); Dietary Supplement: Placebo comparator (protein)
- Low salt, normal protein treatment period (Other): Placebo / 40 grams of protein daily
  Interventions: Dietary Supplement: Protein; Dietary Supplement: Placebo comparator (salt)

INTERVENTIONS:
Dietary Supplement: Sodiumchloride — Subjects will receive 4 capsules containting 750 NaCl each 2dd, making a total of 6 grams NaCl per day.
  Arms: Normal salt, low protein treatment period; Normal salt, normal protein treatment period
Dietary Supplement: Protein — Subjects will receive 2dd 40 ml of a protein beverage containing 0.5 grams of protein per ml, making a total of 40 grams of protein per day.
  Arms: Low salt, normal protein treatment period; Normal salt, normal protein treatment period
Dietary Supplement: Placebo comparator (salt) — Subjects will receive 4 placebo capsules (identical to salt capsules) 2dd.
  Arms: Low salt, low protein treatment period; Low salt, normal protein treatment period
Dietary Supplement: Placebo comparator (protein) — Subjects will receive 2dd 40 ml of placebo beverage (identical to protein beverage).
  Arms: Low salt, low protein treatment period; Normal salt, low protein treatment period

SUMMARY:
This study evaluates the effect of regulating salt and protein intake on urinevolume in patients with ADPKD treated with a vasopressine V2 receptor antagonist (V2RA). The investigators hypothesize that changing sodium and protein intake will reduce V2RA-induced polyuria.

DETAILED DESCRIPTION:
Autosomal Dominant Polycystic Kidney Disease (ADPKD) is characterized by the formation of numerous cysts in both kidneys and progressive renal function decline leading to renal replacement therapy (RRT) at a median age of 58 years. The first (and at the moment only) drug to slow down renal function decline, is a vasopressin V2 receptor antagonist (V2RA). This medicament slows renal function decline by 26 to 34%. V2RA also causes aquaresis associated side-effects such as polyuria of >6 liter per day in the majority of patients. These side-effects limit wide spread use among ADPKD-patients. Therefore, there is a need to improve its tolerability. While using a V2RA, urine concentrating ability is strongly diminished. Therefore, urine volume is largely determined by total osmolar excretion. This is a well-known fact in nephrogenic diabetes insipidus, a disease with clear pathophysiological similarities to treatment with a vasopressin V2 receptor antagonist (a defect receptor versus pharmacological blockade). A recent study found osmolar excretion to be associated with urinary volume during V2RA treatment. Whether a change in osmolar load changes polyuria during V2RA has not yet been investigated. The investigators hypothesize that changing sodium and protein intake will reduce polyuria.

ELIGIBILITY:
Inclusion criteria:

1. Diagnosis of ADPKD (ravine criteria/documented by nephrologist)
2. Stable treatment regimen of tolvaptan as part of routine clinical care in the highest dose tolerable (preferably 120 mg daily), with a urine osmolality lower than 250 mosmol/L.
3. Age >= 18 years.
4. eGFR >30 ml/min/1.73m2.
5. Providing informed consent.
6. Compliance to the recommended diet at two consecutive times.

Exclusion criteria:

1. Patients who, in the opinion of the investigator may present a safety risk.
2. Patients who are unlikely to adequately comply to the trial's procedures (due for instance to medical conditions likely to require interruption or discontinuation, history of substance abuse or non-compliance).
3. a. Patients taking medication likely to confound endpoint assessments:

   * lithium in any dosing regimen;
   * chronic use of systemic corticosteroids in any dosage;
   * chronic use of any diuretics in any dosing regimen;
   * daily use of any NSAIDs in any dosing regimen;

3. b. Patients having concomitant illnesses likely to confound endpoint assessments (e.g. diabetes mellitus for which medication is needed or diabetes insipidus).

4. Women who are pregnant or breastfeeding. 5. Patients with a blood pressure over 160/100 mm Hg at baseline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2020-09-07 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
24-hour urine volume | Baseline, week 2, week 4, week 6, week 8.
  Change in 24-hour urine volume as percentage, comparing the mean of the volumes collected during baseline with the mean of the two volumes collected at the end of each treatment period.

SECONDARY OUTCOMES:
Serum copeptin levels | Baseline, week 2, week 4, week 6, week 8.
  Change in serum copeptin levels, comparing copeptin level measured at baseline with copeptin level measured at the end of each treatment period.
mGFR | Baseline, week 2, week 4, week 6, week 8.
  Change in measured GFR, comparing mGFR measured at baseline with mGFR measured at the end of each treatment period.
Blood pressure | Baseline, week 2, week 4, week 6, week 8.
  Change in blood pressure, comparing blood pressure measured at baseline with blood pressure measured at the end of each treatment period.
Quality of life, assesed by using the ADPKD-IS questionnaire. | Baseline, week 2, week 4, week 6, week 8.
  Change in reported quality of life, comparing reported quality of life at baseline to reported quality of life at the end of each treatment period. To assess quality of life, the ADPKD-IS questionnaires will be used.
Quality of life, assesed by using the NADIQ-questionnaire. | Baseline, week 2, week 4, week 6, week 8.
  Change in reported quality of life, comparing reporter quality of life at baseline to reported quality of life at the end of each treatment period. To assess quality of life, the NADIQ-questionnaires will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Esther Meijer, Dr., Principal Investigator — Universitar Medical Centre Groningen
Locations (1):
- UMC Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] St Pierre K, Cashmore BA, Bolignano D, Zoccali C, Ruospo M, Craig JC, Strippoli GF, Mallett AJ, Green SC, Tunnicliffe DJ. Interventions for preventing the progression of autosomal dominant polycystic kidney disease. Cochrane Database Syst Rev. 2024 Oct 2;10(10):CD010294. doi: 10.1002/14651858.CD010294.pub3. PMID 39356039